CLINICAL TRIAL: NCT06576024
Title: Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in HIV-infected People Aged 1-50 Years: A Phase IV Clinical Trial
Brief Title: Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in HIV-infected People
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LiuZhou People's Hospital (Other)
Collaborators: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Zhongsheng Jiang, Chief physician, LiuZhou People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023010-HAVMHYM(IIT)
Record Dates: First submitted 2024-03-20; First posted 2024-08-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis A; Immunodeficiency; HIV Infections
MeSH Terms: conditions — Hepatitis A; Immunologic Deficiency Syndromes; HIV Infections | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Intervention Model Description: This study aims to evaluate the immunogenicity and safety of hepatitis A vaccine in HIV-infected people, thus the vaccine is considered to be a kind of intervention. We divided HIV-infected people into different groups according to their HIV virus loads to make comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants aged 1-17 years old (Experimental): Participants aged 1-17 years old in the immunogenicity and safety study
  Interventions: Biological: 2 doses of HAV
- HAV susceptible participants aged 18-50 years old (Experimental): HAV susceptible participants aged 18-50 years old in the immunogenicity and safety study
  Interventions: Biological: 2 doses of HAV
- HAV unsusceptible participants aged 18-50 years old (Experimental): HAV unsusceptible participants aged 18-50 years old in the immunogenicity and safety study
  Interventions: Biological: 2 doses of HAV
- Other participants aged 18-50 years old (Experimental): Other participants aged 18-50 years old in the safety study
  Interventions: Biological: At least one dose of HAV

INTERVENTIONS:
Biological: 2 doses of HAV — Participants will receive two doses of HAV with a 6-month interval
  Arms: HAV susceptible participants aged 18-50 years old; HAV unsusceptible participants aged 18-50 years old; Participants aged 1-17 years old
Biological: At least one dose of HAV — Participants will receive the first dose of HAV and willreceive the second dose with a 6 -month interval voluntarily.
  Arms: Other participants aged 18-50 years old

SUMMARY:
Approximately 400 HIV-infected participants aged 1-50 years old will be recruited according to the inclusion and exclusion criteria. Among them, more than 180 participants will be recruited in the immunogenicity and safety study. Each of them will receive 2 doses of the HAV vaccine with a 6-month interval. Blood samples will be drawn before and 1 month after each dose to detect the HAV antibodies to evaluate the immunogenicity of the vaccines. Other people will be recruited in the safety study and receive at least one dose of the HAV vaccine. All the participants will report the adverse events within one month after each dose.

DETAILED DESCRIPTION:
Approximately 400 HIV-infected participants aged 1-50 years old will be recruited in terms of inclusion and exclusion criteria. All participants will receive one dose of the hepatitis A vaccine and have their blood and urine samples collected before and after vaccination for laboratory-related indicator testing. At least 120 HAV-susceptible participants (with anti-HAV antibodies negative before vaccination) and 60 HAV-unsusceptible participants (with anti-HAV antibodies positive before vaccination) aged 18-50 years old, and an unlimited number of HIV-infected children aged 1-17 years old will be included into immunogenicity study, with rest participants included into safety study. Participants in immunogenicity study will receive the second dose of hepatitis A vaccination with a 6-month interval. Blood and urine samples will be collected 1 month, 6months (before second vaccination), and 7 months (1month after second vaccination) after the first vaccination. Participants in safety study will receive second vaccination voluntarily. Adverse events in both immunogenicity and safety study will be collected within 30 days after each dose of vaccination using smartphone mini program or diary cards.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected participants aged 1-50 years old
* The HIV viral loads of participants in the past 12 months were supposed to be less than 200 copies/ml
* Participants or his/her guardian can fully understand and voluntarily sign the informed consent 4. Participants who are willing to participate in the 7-month follow-up 5. Participants who can provide valid legal identification

Exclusion Criteria:

* Participants who have infected with hepatitis A;
* Participants who have been vaccinated with inactivated or live-attenuated hepatitis A vaccine, or hepatitis A and B combined vaccine
* Participants who are allergic constitution or severe allergic to vaccines or components in the past (such as acute allergic reaction, angioedema, dyspnea, etc.)
* Pregnant women and lactating women
* People suffering from uncontrolled epilepsy and other serious neurological diseases (such as transverse myelitis, Guillain-Barré syndrome, demyelinating diseases, etc.)
* Participants with fever (axillary temperature ≥37.3℃) during vaccination, or acute exacerbation of chronic diseases, or participants with uncontrolled severe chronic diseases, or suffering from acute diseases
* Participants who have received other experimental drugs within 30 days before vaccination with the experimental vaccine
* Participants who have received live-attenuated vaccine withins 14 days before vaccination with the experimental vaccine
* Participants who have received subunit or inactivated vaccines within 7 days before vaccination with experimental vaccine
* According to the investigator's judgment, participants who has any other factors that make him or her unsuitable for vaccination

Exclusion Criteria of second vaccination:

Participants who meet one of the following events (1) to (4), should not receive the second vaccination, but can continue other study steps according to the investigator's judgment; if participants who meet one of the following events (5) or (6), can still receive the second vaccination according to the investigator's judgment.

Participants who meet one of the following events (7) to (10) can postponed the second vaccination within the time window specified in the protocal.

1. Vaccines of the same type other than the experimental vaccine were used during the study;
2. Any serious adverse reaction that is causally related to the experimental vaccination
3. Severe allergic reaction or hypersensitivity reaction after vaccination (including urticaria/rash occurring within 30 minutes after vaccination)
4. Pregnant after the first vaccination (those who had positive result for urine pregnancy test or those who are known to be pregnant)
5. Acute or recently diagnosed chronic disease that occurred after the first vaccination
6. Other reactions (including severe pain, severe swelling, severe limitation of activity, persistent high fever, severe headache, or other systemic or local reactions) are diagonosed by investigator
7. Suffering from acute illness (acute illness refers to moderate or severe illness with or without fever);
8. Axillary temperature ≥37.3℃ during vaccination;
9. Have received subunit vaccine or inactivated vaccine within 7 days, and have received live attenuated vaccine within 14 days
10. According to the investigator's judgment, participants who has any other factors that make him or her unsuitable for vaccination

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 392 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of anti-HAV antibodies 30 days after 2 doses of hepatitis A vaccination among HIV-infected participants with hepatitis A susceptibility | 30 days after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Incidences of adverse reactions within 30 days after each dose of hepatitis A vaccination | 0-30 days after each dose of hepatitis A vaccination
  safety evaluation

SECONDARY OUTCOMES:
GMCs of anti-HAV antibodies 30 days after 2 doses of hepatitis A vaccination among HIV-infected participants with hepatitis A susceptibility | 30 days after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
GMIs of anti-HAV antibodies 30 days after 2 doses of hepatitis A vaccination among HIV-infected participants with hepatitis A susceptibility | 30 days after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Seropositive rates of anti-HAV antibodies 30 days after 2 doses of hepatitis A vaccination among HIV-infected participants with hepatitis A susceptibility | 30 days after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Seroconversion rates of anti-HAV antibodies 30 days and 6 months after the first dose of hepatitis A vaccination among HIV-infected participants with hepatitis A susceptibility | 30 days and 6 months after one dose of hepatitis A vaccination
  Immunogenicity evaluation
Seropositive rates of anti-HAV antibodies 30 days and 6 months after 1 dose of hepatitis A vaccination among HIV-infected participants without hepatitis A susceptibility | 30 days and 6 months after 1 dose of hepatitis A vaccination
  Immunogenicity evaluation
GMCs of anti-HAV antibodies 30 days and 6 months after 1 dose of hepatitis A vaccination among HIV-infected participants without hepatitis A susceptibility | 30 days and 6 months after 1 dose of hepatitis A vaccination
  Immunogenicity evaluation
GMIs of anti-HAV antibodies 30 days and 6 months after 1 dose of hepatitis A vaccination among HIV-infected participants without hepatitis A susceptibility | 30 days and 6 months after 1 dose of hepatitis A vaccination
  Immunogenicity evaluation
Incidences of adverse reactions within 7 days after each dose of hepatitis A | 0-7 days after each dose of hepatitis A vaccination
  safety evaluation
Incidences of adverse events within 7 days and within 30 days after each dose of hepatitis A vaccination | 0-7 days and 0-30 days after each dose of hepatitis A vaccination
  safety evaluation
Seroconversion rates of anti-HAV antibodies 30 days after 1 does, 30 days and 6 months after 2 doses of hepatitis A vaccination among HIV-infected participants with anti-HAV antibodies seropositivity | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Seropositive rates of anti-HAV antibodies 30 days after 1 does, 30 days and 6 months after 2 doses of hepatitis A vaccination among HIV-infected participants with anti-HAV antibodies seropositivity | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
GMC of anti-HAV antibodies 30 days after 1 does, 30 days and 6 months after 2 doses of hepatitis A vaccination among HIV-infected participants with anti-HAV antibodies seropositivity | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
GMIs of anti-HAV antibodies 30 days after 1 does, 30 days and 6 months after 2 doses of hepatitis A vaccination among HIV-infected participants with anti-HAV antibodies seropositivity | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
The difference in virus loads of HIV before and after vaccination among HIV-infected people | before and within 1 year after vaccination
  safety evaluation

OTHER OUTCOMES:
Correlation of T-lymphocyte levels with the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of virus titers of HIV with the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of age with the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of hepatitis B co-infection with the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of hepatitis C co-infection with the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of ALT levels with the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of AST levelswith the pre-vacciantion hepatitis A antibodies GMCs | before vaccination
  Immunogenicity evaluation
Correlation of T lymphocyte levels with the pre-vacciantion seropositivity rates of hepatitis A antibodies | before vaccination
  Immunogenicity evaluation
Correlation of virus titers with the pre-vacciantion seropositivity rates of hepatitis A antibodies | before vaccination
  Immunogenicity evaluation
Correlation of age with the pre-vacciantion seropositivity rates of hepatitis A antibodies | before vaccination
  Immunogenicity evaluation
Correlation of hepatitis B co-infection with the pre-vacciantion seropositivity rates of hepatitis A | before vaccination
  Immunogenicity evaluation
Correlation of hepatitis C co-infection with the pre-vacciantion seropositivity rates of hepatitis A | before vaccination
  Immunogenicity evaluation
Correlation of ALT levels with the pre-vacciantion seropositivity rates of hepatitis A antibodies | before vaccination
  Immunogenicity evaluation
Correlation of AST levels with the pre-vacciantion seropositivity rates of hepatitis A antibodies | before vaccination
  Immunogenicity evaluation
Correlation of T-lymphocyte levels with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of virus titers of HIV with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of age with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis B co-infection with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis C co-infection with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of ALT levels with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of AST levels with the post-vacciantion hepatitis A antibodies GMCs | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of T-lymphocyte levels with the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of virus titers of HIV with the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of age with the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis B co-infectionwith the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis C co-infectionwith the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of ALT levels with the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of AST levels with the post-vacciantion seropositivity rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of T-lymphocyte levels with the GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of virus titers of HIV with GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of age with the GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis B co-infection with GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis C co-infection with GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of ALT levels with the GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of AST levels with the GMIs of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of T-lymphocyte levels seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of virus titers of HIV with seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of age with seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis B co-infection with seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of hepatitis C co-infection with seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of ALT levels with seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation
Correlation of AST levels with seroconversion rates of hepatitis A antibodies | 30 days after 1 dose, 30 days and 6 months after 2 doses of hepatitis A vaccination
  Immunogenicity evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Liuzhou People's Hospital, Liuchow, Guangxi, China